CLINICAL TRIAL: NCT02158442
Title: Randomized Study Comparing Clinical and Microbiological Efficacy of Timentin Delivered Via Percutaneous Isolated Limb Perfusion (PILP) or Intravenous Infusion in Diabetic Subjects With Moderate to Severe Lower Limb Infection
Brief Title: Technology That Permits Focal Dose of Antibiotics to be Delivered to Lower Limb(s) of Diabetic Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Osprey Medical, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: O-PILP-C01 - Part B
Record Dates: First submitted 2014-04-11; First posted 2014-06-06 (Estimated); Results first posted 2016-08-03 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-08

CONDITIONS: Diabetes; Infection
Keywords: Diabetes; Lower limb infection; Significant wound infections; Intravenous antibiotics; Timentin
MeSH Terms: conditions — Diabetes Mellitus; Infections | interventions — Parturition; ticarcillin-clavulanic acid; Ticarcillin; Clavulanic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Group (Experimental): The Treatment Group received intravenous Timentin prior to their PILP procedure.
  Interventions: Procedure: Percutaneous Isolated Limb Perfusion (PILP) delivery; Drug: Timentin
- Control Group (Active Comparator): The Control Group received standard dosings of intravenous Timentin plus other standard care.
  Interventions: Drug: Timentin

INTERVENTIONS:
Procedure: Percutaneous Isolated Limb Perfusion (PILP) delivery — The Percutaneous Isolated Limb Perfusion (PILP) delivery intervention procedure enables the use of existing antibiotic therapies in a more targeted and aggressive fashion; it addresses limitations associated with the use of conventional antibiotic drug delivery. As part of the procedure, the circulation of the limb is isolated separately from the general circulatory system enabling the delivery of antibiotic at high therapeutic doses that are not achievable when standard doses are administered intravenously.
  Arms: Treatment Group
Drug: Timentin — The Control Group will receive standard dosings of intravenous Timentin plus other standard care.
  Other Names: Ticarcillin and Clavulanate

SUMMARY:
The use of the Percutaneous Isolated Limb Procedure (PILP) which enables the use of existing antibiotic therapies in a more targeted and concentrated fashion in patients with diabetes who have a significant lower limb infection and it is deemed that IV antibiotics are needed in order to salvage the limb or life.

DETAILED DESCRIPTION:
During the PILP procedure, the circulation of the limb is isolated separately from the general circulatory system thereby enabling the delivery of antibiotics only to the limb. Limb isolation is achieved by creating an "artificial" circuit where catheters are inserted into the major artery and vein of the lower limb.

ELIGIBILITY:
Inclusion Criteria:

* M or F subjects 18 - 90 years old
* Subject has pre-existing diabetes diagnosis
* Subject has significant infection below the ankle of soft tissue and may include bone, and IV antibiotics are needed in order to salve limb or life
* Consequence of infected wound would require Std of Care share debridement
* Subject willing and able to provide written informed consent
* Subject willing and able to comply with requirements of study protocol including pre-defined follow-up evaluations
* PROCEDURAL INCLUSION CRITERIA: successful cannulation of the femoral artery and vein and placement of the venous support device

Exclusion Criteria:

* Allergy to contrast media
* Known bleeding disorder including thrombocytopenia
* Recent AMI or elevated Troponin levels within last 30 days
* Penicillin sensitivity; Timentin sensitivity
* Female subjects known to be or suspected to be pregnant or lactating
* Subject unable to comply with instructions; especially to remain supine for duration of recirculation procedure
* Subjects who have participated in any other clinical trial or taken investigational drug within 30 days of study enrollment
* The PI determines the subject is not an appropriate subject for the study
* PROCEDURAL EXCLUSION CRITERIA: Subjects anatomy interferes with or is expected to prohibit successful cannulation of the femoral vessels or placement of the venous support device
* Known severe proximal femoral artery vascular disease precluding placement of perfusion catheters

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-10; Primary Completion 2015-02 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Wraight, Assoc. Prof., Principal Investigator — Royal Melbourne Hospital, Head, Diabetic Foot Unit
Locations (1):
- Royal Melbourne Hospital, Parkville, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject enrolled 17 Oct 2013. Study completion 28 Feb 2015.
Period: Overall Study
Arm/Group | Treatment Group | Control Group
Started | 8 | 7
Completed | 6 | 7
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Perfusion staff not available | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group | Control Group | Total
Number analyzed (Participants) | 6 | 7 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 7
  >=65 years | 2 | 4 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.2 (8.3) | 63.0 (5.9) | 63.5 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 6 | 7 | 13
Region of Enrollment [Number; unit: participants]
  Australia | 6 | 7 | 13

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Timentin Delivered by PILP Procedure (Treatment Group) Versus Intravenous Delivery (Control Group) at Reducing Microbiological Load in Subjects With Diabetes, and Significant Wound Infection of the Lower Limb.
Description: Reduction in microbiological load, including assessment of CFU, infection type and antibiotic sensitivity between the two groups over time. To compare the efficacy of Timentin delivered by PILP procedure (Treatment Group) versus intravenous delivery (Control Group) at reducing microbiological load in subjects with diabetes, and significant wound infection of the lower limb.
Time Frame: Day 3
Population: Treatment Group: 5 of the 5 analyzable microbiological loads resulted in a reduction. 1 was not analyzable.
  Control Group: 3 of the 3 analyzable microbiological loads resulted in a reduction. 4 were not analyzable.
Measure: Number; unit: participants
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 5 | 3
participants | 5 | 3

ADVERSE EVENTS:
Time Frame: Through 28 days.
Arm/Group | Treatment Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/7
Other Adverse Events (participants affected / at risk) | 0/6 | 0/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=6) | Control Group (N=7)
MCA Infarct (Cardiac disorders) | 0 (0) | 1 (1) — R MCA Infarct on control subject

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No